CLINICAL TRIAL: NCT05524168
Title: SBRT Combined With Programmed Death 1 (PD-1) Antibody and Chemotherapy in Nasopharyngeal Carcinoma With Oligometastasis: A Prospective, Multicenter, Single-arm, Phase II Clinical Trial
Brief Title: SBRT Combined With PD-1 Antibody and Chemotherapy in Oligometastatic Nasopharyngeal Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Shenzhen People's Hospital (Other); First People's Hospital of Foshan (Other); Jiangxi Provincial Cancer Hospital (Other); The First Affiliated Hospital of Xiamen University (Other); Chongqing University Cancer Hospital (Other)
Responsible Party: Principal Investigator, Zhao Chong, Dr. Prof., Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SBRT+PD-1+Chemo for mNPC
Record Dates: First submitted 2022-08-29; First posted 2022-09-01 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: SBRT; PD-1 antibody; Chemotherapy; Efficacy; Safety; Oligometastasis
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — camrelizumab; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT+PD-1+Chemotherapy (Experimental): Patients will receive SBRT first, then PD-1 antibody (Camrelizumab 200mg/Q3W) and chemotherapy (cisplatin 80mg/m2 on d1, gemcitabine 1000mg/m2, d1 and d8, Q3W, maximum 6 cycles), followed by Camrelizumab (200mg/Q3W) until progressive disease, intolerable toxicity, withdrawal of consent or a maximum of 1 year treatment.
  Interventions: Radiation: SBRT; Drug: Camrelizumab; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Radiation: SBRT — SBRT for metastatic lesions
Drug: Camrelizumab — Maximum 6 cycles for combined therapy. Camrelizumab maintenance for 1 year.
  Other Names: SHR-1210
Drug: Gemcitabine — Maximum 6 cycles for combined therapy.
Drug: Cisplatin — Maximum 6 cycles for combined therapy.

SUMMARY:
This is a multicenter, single-arm, phase II clinical trial. The purpose of this study is to evaluate the efficacy and adverse effect of SBRT combined with programmed death 1 (PD-1) antibody and chemotherapy in nasopharyngeal carcinoma patients with oligometastasis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as metastatic NPC with no more than 5 metastatic lesions;
* Histopathological diagnosis of NPC;
* ECOG 0-1 point;
* Has not received prior systemic treatment, such as radiotherapy, chemotherapy, immunotherapy or biotherapy;
* No contraindications to immunotherapy and chemoradiotherapy;
* Every metastatic lesions could receive SBRT safely;
* Subject must have a measurable target lesion based on RECIST v1.1;
* Adequate marrow function: WBC count ≥ 3×10E9/L, NE count ≥ 1.5×10E9/L, HGB ≥ 90g/L, PLT count ≥ 100×10E9/L;
* Adequate liver function: ALT/AST ≤ 2.5×ULN, TBIL ≤ 2.0×ULN;
* Adequate renal function: BUN/CRE ≤ 1.5×ULN or endogenous creatinine clearance ≥ 60ml/min (Cockcroft-Gault formula);
* Take effective contraceptions during and three months after treatment;
* Patients must be informed of the investigational nature of this study and give written informed consent.

Exclusion Criteria:

* Allergic to monoclonal antibodies, any PD-1 antibody components, gemcitabine and cisplatin;
* Unexplained fever > 38.5 ℃, except for tumor fever;
* Have active autoimmune disease (e.g., uveitis, enteritis, hepatitis, hypophysitis, nephritis, vasculitis, hyperthyroidism, and asthma requiring bronchodilator therapy);
* Have a known history of human immunodeficiency virus (HIV), active Hepatitis B (HBV-DNA ≥10E3copiers/ml) or hepatitis C virus (HCV) antibody positive;
* Have previously treated with PD-1 antibody or other immunotherapy for PD-1/PD-L1 pathway;
* Have New York Heart Association (NYHA) class 3 or 4, unstable angina, myocardial -infarction within 1 year, or clinically meaningful arrhythmia that requires treatment; Have known allergy to large molecule protein products or any compound of study therapy;
* Pregnant or breastfeeding;
* Prior malignancy except adequately treated non-melanoma skin cancer, in situ cervical cancer, and papillary thyroid carcinoma;
* Have received a live vaccine within 30 days of planned start of study therapy Has psychiatric drug or substance abuse disorders that would interfere with cooperation with the requirements of the trial;
* Any other condition, including mental illness or domestic/social factors, deemed by the investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interferes with the interpretation of the results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2022-11-25 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | up to 12 months
  Defined as the time from randomization to the first occurrence of disease progression as determined according to RECIST v1.1 or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival | up to 12 months
  Defined as the time from randomization to death from any cause.
Objective Response Rate | up to 12 months
  The percentage of patients with CR and PR assessed according to RECIST v1.1.
Disease Control Rate | up to 12 months
  The proportion of patients who have achieved complete response, partial response and stable disease according to RECIST v1.1.
Adverse Events | up to 12 months
  All adverse event or serious adverse event that occurred during the study period according to CTCAE v 4.03
QoL | up to 12 months
  Assessed by EQ-5D-5L questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Chong Zhao, MD. PhD., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China